CLINICAL TRIAL: NCT04186494
Title: The Benefit of a Liraglutide-based Weight Management Alone or in Addition to Standard CPAP Therapy on Metabolic Function in Patients With Obstructive Sleep Apnoea (OSA) - an Explorative, Proof-of-concept Study
Brief Title: Effect of Liraglutide vs CPAP on Cardiometabolic Outcomes in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's University Hospital, Ireland (Other)
Collaborators: University College Dublin (Other); Health Research Board, Ireland (Other)
Responsible Party: Principal Investigator, Dr Silke Ryan, Associate Professor, Consultant in Respiratory and Sleep Medicine, St Vincent's University Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RS19-023
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Liraglutide; Continuous positive airway pressure; Insulin resistance; Vascular inflammation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Insulin Resistance | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous positive airway pressure (CPAP) (Active Comparator): Standard CPAP Therapy
  Interventions: Device: Continuous positive airway pressure treatment
- Liraglutide-based weight loss regimen (Experimental): Once daily s.c. injections of Liraglutide, starting at a dose of 0.6 mg with weekly 0.6 mg increments to 3.0 mg in adjunct to advice on a weight-reduction diet and physical exercise
  Interventions: Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml
- Combination CPAP/Liraglutide (Experimental): Combination of both interventions
  Interventions: Combination Product: Liraglutide and CPAP

INTERVENTIONS:
Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml — GLP-1 analogue treatment in combination with advice on diet and physical exercise
  Arms: Liraglutide-based weight loss regimen
Device: Continuous positive airway pressure treatment — Gold standard treatment for obstructive sleep apnea
  Arms: Continuous positive airway pressure (CPAP)
Combination Product: Liraglutide and CPAP — Combination of both treatments
  Arms: Combination CPAP/Liraglutide

SUMMARY:
This is an explorative, proof-of-concept study exploring the potential therapeutic role of a Liraglutide-based weight loss regimen versus standard CPAP or the combination of both on metabolic parameters, blood pressure, endothelial function, coronary artery calcification, vascular inflammation and apnea/hypopnea index in non-diabetic patients with moderate to severe obstructive sleep apnea

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed moderate-severe OSA (by standard PSG)
* Body mass index between 30 - 40
* Age 18 - 60 years
* Able to provide written, informed consent

Exclusion Criteria:

* Pregnancy
* Requirement for supplemental oxygen
* Previous diagnosis of OSA or previous CPAP treatment
* Diagnosis of Diabetes
* Previous treatment with GLP-1 analogue
* Previous surgical treatment for obesity
* Active treatment for malignancy or severe psychiatric disorder
* Acute coronary syndrome or stroke within 3 months prior to study
* History of decompensated heart failure
* Professional drivers or drivers with a history of road-traffic accident due to sleepiness
* Severe excessive daytime sleepiness defined as Epworth sleepiness scale >15

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 6 months
  Improvement in insulin resistance defined by HOMA-IR

SECONDARY OUTCOMES:
Weight | 6 months
  Change in body mass index
Glucose tolerance | 6 months
  Change in glucose tolerance measured by oral glucose tolerance test
OSA Severity | 6 months
  Change in apnea/hypopnea index as per polysomnography
Blood pressure | 6 months
  Change in 24-hour blood pressure
Endothelial function | 6 months
  Change in microvascular endothelial function measured by EndoPat
Coronary artery calcification | 6 months
  Change in coronary artery calcification score determined by Coronary artery CT
Vascular inflammation | 6 months
  Change in vascular inflammation determined via FDG-PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Silke Ryan, PhD, MD, Principal Investigator — St Vincent's University Hospital, University College Dublin
Locations (1):
- St Vincent's University Hospital, Dublin, Dublin 4, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Donnell C, Crilly S, O'Mahony A, O'Riordan B, Traynor M, Gitau R, McDonald K, Ledwidge M, O'Shea D, Murphy DJ, Dodd JD, Ryan S. Continuous Positive Airway Pressure but Not GLP1-mediated Weight Loss Improves Early Cardiovascular Disease in Obstructive Sleep Apnea: A Randomized Proof-of-Concept Study. Ann Am Thorac Soc. 2024 Mar;21(3):464-473. doi: 10.1513/AnnalsATS.202309-821OC. PMID 38096106